CLINICAL TRIAL: NCT02482506
Title: BRE-WL4AA Moving Forward: A Weight Loss Intervention for African-American Breast Cancer Survivors
Brief Title: Moving Forward: A Weight Loss Intervention for African-American Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: University of Chicago (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Melinda Stolley, Associate Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: BRE-WL4AA
Record Dates: First submitted 2015-04-30; First posted 2015-06-26 (Estimated); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Breast Cancer
Keywords: African American; Overweight; Adults
MeSH Terms: conditions — Breast Neoplasms; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SG-WLP (Other): Self-guided weight loss program
  Interventions: Behavioral: SG-WLP
- MF-WLP (Active Comparator): Moving Forward Weight Loss Program
  Interventions: Behavioral: MF-WLP

INTERVENTIONS:
Behavioral: MF-WLP — The first meeting each week includes a 60-minute class that addresses health knowledge, attitudes, and self-monitoring of weight, food and physical activity; realistic goal setting; stimulus control; problem solving; cognitive restructuring and relapse prevention. Other class activities include weekly weigh-in; increasing awareness of portions by weighing and measuring foods; creating stimulus control plans for home, car and work; identifying barriers to healthy eating and/or exercise; going on a field trip to a local grocery store to practice reading food labels; creating an eating out management plan; and identifying high risk situations and brainstorming ways to manage them. This meeting also includes a 60-minute exercise class. The second meeting each week is a stand-alone 60-minute exercise class that will incorporate a variety of activities. A one-year CPD fitness club membership and home exercise DVDs will be provided.
  Other Names: Moving Forward Guided Weight Loss Program
  Arms: MF-WLP
Behavioral: SG-WLP — Control participants will be provided with a 24-week weight loss curriculum; this includes a binder with their personal daily caloric recommendation, all intervention handouts, a copy caloric guidelines and useful weight loss tools. Upon randomization, each control participant will be introduced to the program materials and encouraged to tailor the weight loss program for themselves. The study team will call each control participant once a month during this 6-month program period to check in. In addition, after the follow-up data collection, control participants will receive a one-year membership to the CPD fitness center.
  Other Names: Self-guided Weight Loss Program
  Arms: SG-WLP

SUMMARY:
This is a randomized intervention study to examine the effects of the Moving Forward Guided Weigh Loss Intervention compared to a self-guided weight loss program on BMI and behavioral, biological, and psychosocial outcomes in overweight and obese African American women diagnosed with Stage I, II, or III breast cancer.

DETAILED DESCRIPTION:
This is a randomized study with 300 African American (AA) breast cancer survivors to be conducted in Chicago Park District (CPD) facilities. The study will be based in six predominantly AA communities in Chicago (Roseland, Pullman, Englewood, Chatham, Austin, South Shore, Woodlawn, Calumet Heights, North Lawndale and Grand Crossing). These communities have at least one CPD fitness center, have populations that are at least 90% or more AA and have similar socioeconomic statuses. Fifty AA breast cancer survivors will be recruited from each community (25 treatment/ 25 control).

The Moving Forward intervention integrates concepts from Social Cognitive Theory (SCT) and the Socio-Ecological Model (SEM) to promote independent behavior change. SCT suggests that behavior can be explained by the dynamic interaction between behavior, personal factors (e.g., self-efficacy), and the environment (e.g, social support). Self-efficacy is a person's confidence in performing a particular behavior and overcoming barriers to that behavior. A number of studies have supported the mediating role of self-efficacy in making independent health behavior changes.

The overall goal of Moving Forward is to make independent changes in health behaviors to promote a healthy weight. The weight loss goal will be consistent with the recommendations of an expert panel at National Institutes of Health (NIH). Dietary goals aimed at producing weight loss, decreasing BC recurrence risk, and improving overall health include 1) a decrease in daily caloric intake (based on weight in pounds X 12 kcal/day with 500-750 calories subtracted to create an energy deficit); 2) a decrease in dietary fat consumption to 20% of total calories; 3) an increase in fruit and vegetable consumption to 7 daily servings; and 4) an increase in fiber to 25 grams per day. For exercise, participants will gradually increase their activity to a minimum of 180 minutes per week at 55-65% maximal heart rate.

ELIGIBILITY:
Inclusion Criteria:

* Self-identification as Black or African American (including individuals who are bi-racial but identify themselves as Black or AA)
* Female
* Stage I, II, and III invasive breast carcinoma
* Treatment (surgery, chemotherapy and/or radiation) completed at least 6 months prior to recruitment (ongoing treatment with tamoxifen or AIs is acceptable)
* Age 18 or above at time of diagnosis
* BMI at least 25 km/m2
* Physically able to participate in a moderate physical activity program as assessed by a screening questionnaire and PCP approval.
* Agreeable to random assignment and data collection including blood draw.
* Able to attend twic weekly classes for 6 months.

Exclusion Criteria:

* Plans to move from the community during the study
* Medical condition limiting adherence as assessed by PCP
* History of significant mental illness
* Currently pregnant, less than 3 months post-partum, or pregnancy anticipated during the study..
* Current/planned use of an FDA-approved or over the counter weight loss medication.
* Participation in another structured weight loss program

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2011-07; Primary Completion 2016-03 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Change in weight | 6 months
  weight in kilograms
change in weight | 12 months
  weight in kilograms

CONTACTS AND LOCATIONS:
Overall Officials: Melinda Stolley, PhD, Principal Investigator — University of Illinois at Chicago

REFERENCES:
- [Derived] Springfield S, Odoms-Young A, Tussing-Humphreys L, Freels S, Stolley M. Adherence to American Cancer Society and American Institute of Cancer Research dietary guidelines in overweight African American breast cancer survivors. J Cancer Surviv. 2019 Apr;13(2):257-268. doi: 10.1007/s11764-019-00748-y. Epub 2019 Apr 13. PMID 30982113
- [Derived] Stolley MR, Sharp LK, Fantuzzi G, Arroyo C, Sheean P, Schiffer L, Campbell R, Gerber B. Study design and protocol for moving forward: a weight loss intervention trial for African-American breast cancer survivors. BMC Cancer. 2015 Dec 29;15:1018. doi: 10.1186/s12885-015-2004-4. PMID 26715447